CLINICAL TRIAL: NCT03119285
Title: Genes Contributing to Hereditary Ovarian Cancer in Women and BRCA1/2 Wildtype Families
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Elizabeth Swisher, Professor, Obstetrics & Gynecology, University of Washington
Other Study IDs: STUDY00001583
Record Dates: First submitted 2016-10-31; First posted 2017-04-18 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; BRCA1; BRCA2; BROCA
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be obtained and constitutional DNA extracted. The investigators will obtain paraffin embedded tumor blocks from enrolled participants.
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators propose to test for non-BRCA1/2 mutations in new and existing families with hereditary ovarian cancer in order to better define penetrance and associated malignancies of rare ovarian cancer susceptibility genes. The hypothesis is at least one third of hereditary ovarian carcinoma families wildtype for BRCA1/2 can be solved using an updated version of BROCA (BROCA-HR) that targets 47 genes, including all known ovarian cancer genes and additional candidate genes in related pathways. The objective is to identify families with mutations in rare ovarian cancer susceptibility genes and test both affected and unaffected family members, thereby generating a rough estimate of penetrance for each mutated gene as well as identify new ovarian cancer susceptibility genes. The investigators also plan to enroll self identified African America women, who have been drastically under-represented in clinical cancer genetic testing programs and in OC susceptibility research.

DETAILED DESCRIPTION:
There is more to hereditary ovarian cancer than the breast and ovarian cancer susceptibility genes BRCA1 and BRCA2 (BRCA1/2). Next generation sequencing techniques have made it possible to sequence multiple candidate ovarian carcinoma susceptibility genes simultaneously. The King Laboratory has developed a targeted capture and massively parallel sequencing test called BROCA to evaluate mutations in known or suspected breast and ovarian cancer genes. In a prospective series of 360 unselected women with ovarian carcinoma, the investigators found that nearly one fourth of women carried mutations in one of 13 genes, and mutations in genes other than BRCA1 and BRCA2 accounted for 26% of all inherited mutations. While BROCA and similar gene panels are already in clinical use, little is known about the relative risks of carrying these non-BRCA1/2 mutations, making it difficult to counsel unaffected family members and develop optimum prevention protocols.

ELIGIBILITY:
Inclusion Criteria:

* ovarian cancer diagnosis with secondary criteria as noted above

Exclusion Criteria:

* age less than 18 yrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will enroll subjects from the following groups:1) African American women with ovarian carcinoma and 2) women with ovarian carcinoma and one of the following criteria:
  1. first or second degree relative with ovarian carcinoma or
  2. developed a second, independent primary invasive cancer or
  3. been identified with a suspected, deleterious, non-BRCA 1/2 mutation
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2013-04; Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Rate of deleterious germline mutations | 10 years
  The rate of deleterious germline mutations in known ovarian cancer genes as identified using BROCA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Swisher, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No